CLINICAL TRIAL: NCT05492318
Title: Open-label, Single-center Study in Healthy Subjects to Investigate the Effect of Oral Givinostat on Pharmacokinetics (PK) of Intravenous and Oral Midazolam and Oral Dabigatran Etexilate (PART 1)
Brief Title: Perpetrator DDI Potential of Givinostat as Inhibitor and Inducer of CYP3A and P-gp Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITF/2357/55 - PART 1; 2021-005756-11 (EudraCT Number)
Record Dates: First submitted 2022-06-09; First posted 2022-08-08 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Drug-Drug Interaction; Heathy Volunteer
Keywords: PK; Pharmacokinetics; Givinostat; Midazolam; Dabigatran
MeSH Terms: interventions — givinostat; givinostat hydrochloride; Midazolam; Dabigatran; Hardness

STUDY DESIGN:
Intervention Model Description: An Open-label, Single-center trial in Healthy Subjects
Masking Description: The study was conducted as open label. Blinding procedures were not applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Givinostat alone or combo with Midazolam IV and with oral Dabigatran, or combo with oral Midazolam (Experimental): On Days 1, 6 and 17, single doses of midazolam 1 mg IV and dabigatran etexilate 75 mg were administered 1 hour after the planned (as per Day 4) morning time of givinostat administration. On Days 2, 7 and 18, a single oral dose of midazolam 2.5 mg oral solution was administered 1 hour after the planned (as per Day 4) morning time of givinostat administration. From Day 4 to Day 18, givinostat 50 mg as oral suspension was administered twice a day, in the morning and in the evening. On Day 19, only the morning dose was administered.
  Interventions: Drug: Givinostat 10 mg/mL; Drug: Midazolam 1mg/ml IV; Drug: Midazolam 2.5 mg oromucosal solution; Drug: Dabigatran etexilate 75 mg oral hard capsules

INTERVENTIONS:
Drug: Givinostat 10 mg/mL — 10 mg/mL oral suspension. Givinostat 10 mg/ml oral suspension was administered once, in the morning, in Days 1, 2, 6, 7, 17 and 18), and twice a day (50 mg as oral suspension), in the morning and in the evening, from the Day 4 to Day 18. On Day 19, only the morning dose was administered.
  Other Names: ITF2357
Drug: Midazolam 1mg/ml IV — Midazolam 1 mg/ml, solution for intravenous administration. Midazolam 1mg/ml IV, single dose, was administered on Days 1, 6 and 17, 1 hour after the planned morning time of givinostat administration. Midazolam IV were administered with the subjects in a semi-recumbent position. Subjects remained semirecumbent until at least 3 hours post-dose.
  Other Names: Aurobindo®
Drug: Midazolam 2.5 mg oromucosal solution — Dose: 2.5 mg oromucosal solution. Midazolam 2.5 mg single oral solution was administered on Days 2, 7 and 18, 1 hour after the planned morning time of givinostat administration.
  Oral midazolam (and dabigatran etexilate) was administered following an overnight fasting of at least 8 hours and subjects remained fasted until at least 3 hours post-dose.
  Oral midazolam (and dabigatran etexilate) was administered with 150 mL of water. Except for water given with the investigational products, no fluids were allowed from 1 hour before midazolam and dabigatran dosing until 2 hours postdose. Water was provided ad libitum at all other times. Midazolam (and dabigatran etexilate) were administered with the subjects in a semi-recumbent position. Subjects remained semirecumbent until at least 3 hours post-dose.
  Other Names: Buccolam®
Drug: Dabigatran etexilate 75 mg oral hard capsules — Dose: 75 mg; Dosage form: hard capsules On Days 1, 6 and 17, dabigatran etexilate 75 mg was administered (with midazolam 1mg IV) 1 hour after the planned morning time of givinostat administration.
  Dabigatran etexilate (and midazolam) was administered following an overnight fasting of at least 8 hours and subjects remained fasted until at least 3 hours post-dose Oral dabigatran etexilate (and oral midazolam) was administered with 150 mL of water. Except for water given with the investigational products, no fluids were allowed from 1 hour before dabigatran (and midazolam) dosing until 2 hours postdose. Water was provided ad libitum at all other times. Dabigatran etexilate (and Midazolam) was administered with the subjects in a semi-recumbent position. Subjects remained semirecumbent until at least 3 hours post-dose.
  Other Names: Pradaxa

SUMMARY:
Primary objective:

1. To assess the potential inhibitory and inducing effect of oral givinostat on the single dose pharmacokinetics (PK) of intravenous or oral midazolam.
2. To assess the potential inhibitory and inducing effect of oral givinostat on the single dose PK of oral dabigatran etexilate.

Secondary objective:

To assess the safety and tolerability of concomitant administration of givinostat plus midazolam and dabigatran etexilate.

DETAILED DESCRIPTION:
This study was planned as a phase I, open-label, 3-part, fixed-sequence, nonrandomized study in healthy male and female subjects. The study evaluated the givinostat (ITF2357) potential drug-drug interaction (DDI) at level of CYP3A-mediated metabolism and P-glycoprotein (P-gp) transport with intravenous or oral midazolam and with oral dabigatran etexilate.

More precisely, the study aimed at assessing the potential (inhibitory or inducing) effect of givinostat on the PK of midazolam IV, on the PK of oral midazolam and on the PK of dabigatran etexilate.

The study lasted from Day 1 to Day 20. Subjects were confined from Day -1 to Day 20. On Days 6 and 17, single doses of 1 mg midazolam IV and 75 mg dabigatran etexilate, were administered 1 hour after the planned morning time of givinostat administration. On day 1, however, drugs were not administered 1h after gininostat.

On Days 7 and 18, a single oral dose of 2.5 mg midazolam oral solution was administered 1 hour after the planned morning time of givinostat administration.

On day 2, however, the drugs were not administered 1h after gininostat.

From Day 4 to Day 18, givinostat 50 mg as oral suspension was administered twice a day, in the morning and in the evening.

On Day 19, only the morning dose was administered.

The following assessments were performed:

* Blood collection for pharmacokinetic analysis on Days 1 to 4, 6 to 9 and 17 to 20.
* Vital signs measurements (BP, PR and RR) on Days 1, 2, and 4 to 19.
* 12-lead ECG on Days 3 to 19.
* Blood collection for laboratory tests (hematology, biochemistry and coagulation on Days 4 and 9 and hematology on Days 6, 12, 15 and 18). Subjects were discharged from BlueClinical Phase I in the morning of Day 20 if allowed by the investigator based on their medical condition. The following procedures were performed:
* Physical examination.
* Collection of body weight.
* Vital signs measurements (BP, PR, RR and body temperature).
* 12-lead ECG.
* Safety laboratory assessments (hematology, biochemistry, coagulation and urinalysis).
* Serum pregnancy test for all female subjects. Subjects returned to the site 10 to 14 days after the end of study to undergo additional assessments as required per protocol.

The total duration of Part 1 for each subject was up to approximately 8 weeks from Screening to Follow-up visit, divided as follows:

* Screening: up to 21 days
* Treatment Period: Days 1 to 20
* Safety follow-up visit: 12±2 days

ELIGIBILITY:
Inclusion criteria

A subject was considered eligible for the study if he/she fulfilled all the inclusion criteria:

1. Subject's written informed consent obtained prior to any study-related procedure.
2. Male or female subject, ≥18 and ≤55 years of age, at the time of signing the informed consent.
3. Body mass index (BMI) of 18.5 to 32.0 kg/m2 inclusive, and body weight ≥55 kg and ≤100 kg for females and body weight ≥60 kg and ≤110 kg for males.
4. Non-smoker or ex-smoker (i.e. someone who abstained from using tobaccoor nicotine-containing products for at least 3 months prior to Screening).
5. No clinically relevant diseases.
6. No major surgery within 4 weeks prior to dosing.
7. No clinically relevant abnormalities on physical examination.
8. No clinically relevant abnormalities on 12-lead ECG.
9. No clinically relevant abnormalities on clinical laboratory tests.
10. Negative test results for anti-Human Immunodeficiency virus 1 and 2 antibodies (anti-HIV-1Ab and anti-HIV-2Ab), Hepatitis B surface antigen (HBsAg) and anti-Hepatitis C virus antibodies (anti-HCVAb).
11. Female subjects are eligible if they are of non-childbearing potential or agree to use a non-hormonal highly effective contraceptive method from 28 days prior to Screening until at least 90 days after the last study drug administration. Nonchildbearing potential female is defined as:

    1. Menopausal, i.e. no menses for ≥ 12 months without an alternative medical cause other than menopause, and a high FSH level.
    2. Pre-menopausal female with documented hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy.

    A non-hormonal effective contraceptive method is defined as:
    1. Intrauterine device.
    2. Bilateral tubal occlusion.
    3. Total abstinence of heterosexual intercourse, in accordance with the lifestyle of the subject.
    4. Vasectomized partner, who has received medical assessment of the surgical success, or clinically diagnosed infertile partner.
12. Male subjects who are sexually active with a female partner of childbearing potential (pregnant or non-pregnant) must use contraception (condom) from investigational product administration up to at least 90 days following the last study drug administration.
13. Male subjects must ensure that his non-pregnant female partner of childbearing potential agrees to consistently and correctly use for the same period a highly effective method of contraception (see Section 8.5.3).
14. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
15. Willingness and capability to comply with the requirements of the study and ability to understand the study procedures and the risks involved.

Exclusion Criteria

A subject was excluded from the study if he/she fulfilled any of the exclusion criteria:

At Screening

1. Previous use of givinostat.
2. History of anaphylaxis reaction or clinically significant drug hypersensitivity reaction (e.g., angioedema, Stevens-Johnson syndrome, acute generalized exanthematous pustulosis, drug-induced hypersensitivity syndrome, druginduced neutropenia).
3. Known history of hypersensitivity and/or allergic reactions to givinostat, histone deacetylases (HDAC) inhibitors or to any excipient in the formulation.
4. History of sorbitol intolerance, sorbitol malabsorption or fructose intolerance.
5. Any medical condition (e.g. gastrointestinal, renal or hepatic, including peptic ulcer, inflammatory bowel disease or pancreatitis) or surgical condition (e.g. cholecystectomy, gastrectomy) that may affect drug pharmacokinetics (absorption, distribution, metabolism or excretion) or subject safety.
6. Systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 60 or over 90 mmHg, or pulse rate lower than 50 or over 100 bpm.
7. QTcF ˃450 msec.
8. Subjects with history of cardiac arrhythmias (documented), family history of sudden cardiac death or history of additional risk factors for torsades-depointes (e.g. heart failure, hypokalemia, long QT syndrome).
9. Having an estimated glomerular filtration (eGFR) < 90 mL/min, based on creatinine clearance calculation by the Cockcroft-Gault formula and normalized to an average surface area of 1.73 m2.
10. Any of the following abnormal laboratory test values:

    1. Platelet count below the lower limit of the normal range (LLN)
    2. Total white blood cells count below the LLN
    3. Hemoglobin below the LLN
    4. Triglycerides above the upper limit of normal range (ULN)
    5. Potassium or magnesium below the LLN
11. Positive urine alcohol, drugs-of-abuse or cotinine screen tests.
12. Positive serum pregnancy test.
13. If woman, she is breast-feeding.
14. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (i.e. more than 14 units of alcohol per week for males or more than 7 units for females).
15. History of drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs [such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives] within 1 year prior to screening.
16. Participation in any clinical trial within the previous 2 months.
17. Participation in more than 2 clinical trials within the previous 12 months.
18. Blood donation or significant blood loss (≥ 450 mL) due to any reason or had plasmapheresis within the previous 2 months.
19. Veins unsuitable for intravenous puncture on either arm.
20. Difficulty in swallowing capsules, tablets or suspensions.
21. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

    Exclusion Criteria:

    At Admission to Treatment Period
22. Any clinically relevant abnormalities on clinical laboratory tests.
23. Positive urine alcohol, drugs-of-abuse or cotinine screen tests.
24. Positive urine pregnancy test.
25. Positive or inconclusive SARS-CoV-2 test prior to admission.
26. Use of prescription or non-prescription medicinal products within the previous 28 days or within 5-half-lives of the medicinal product, whichever is longer.
27. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

    For Part 1 subjects:

    At Screening
28. Known history of hypersensitivity and/or allergic reactions to midazolam, other benzodiazepines, dabigatran etexilate or to any excipient of the formulations.
29. Clinically relevant history of impaired respiratory function, obstructive sleep apnea, myasthenia gravis, respiratory arrest and/or cardiac arrest.
30. History of glaucoma.
31. Presence of respiratory failure.
32. Presence of active clinically significant bleeding.
33. Lesion or condition considered to pose a significant risk factor for major bleeding including, but not limited to: current or recent gastrointestinal ulceration, malignant neoplasms, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities.
34. Presence of a medical condition requiring anticoagulant treatment.

    At Admission to Treatment Period
35. Treatment with anticoagulants within 28 days or 5 drug half-lives, whichever was longer, before admission.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fonseca, MD, Principal Investigator — Blueclinical, Ltd.
Locations (1):
- Hospital da Prelada, 3rd Floor & East Wing 4th Floor Rua Sarmento de Beires, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened between Days -21 to -3 (both inclusive) of study part 1 to confirm that they met the subject selection criteria. Prior to any screening assessment, the Investigator (or an appropriate delegate) obtained informed consent from each subject in accordance with the procedures. 26 subjects were enrolled to study part 1. Please note that the overall figure n=104 is wrong; the system in fact automatically and inappropriately sums up the number of each IMP group.
Groups:
- All Study Participants (SAF and PK Population): Twenty-six (26) subjects (7 women and 19 men) were admitted to study Part 1:
  * single doses of midazolam 1 mg IV + dabigatran etexilate 75 mg were administered 1 hour after the planned morning time of givinostat administration on Days 1, 6 and 17.
  * a single oral dose of midazolam 2.5 mg oral solution was administered 1 hour after the planned morning time of givinostat administration on Days 2, 7 and 18, Please note that From Day 4 to Day 18, givinostat 50 mg as oral suspension was administered twice a day, in the morning and in the evening, while on Day 19 only the morning dose was administered.
  Midazolam and dabigatran etexilate were administered following an overnight fasting of at least 8 hours and subjects remained fasted until at least 3 hours post-dose and were administered with the subjects in a semi-recumbent position. Subjects remained semirecumbent until at least 3 hours post-dose. Oral midazolam and dabigatran etexilate were administered with 150 mL of water. No other fluids were allowed from 1 hour before midazolam and dabigatran dosing until 2 hours postdose.
  Water was provided ad libitum at all other times.
Period: Overall Study
Arm/Group | All Study Participants (SAF and PK Population)
Started | 26
Day 1 - Midazolam (IV) 1 mg + Dabigatran 75 mg (Potential Inhibitory Effect of Givinostat on Midazolam IV and on Dabigatran Analysis Population) | 26
Day 2 - Midazolam (Oral) 2.5 mg (Potential inhibitory effect of Givinostat analysis population) | 26
Days 4-5 - Givinostat 50 mg b.i.d. | 26
Day 6 - Midazolam (IV) 1 mg + Dabigatran 75 mg + Givinostat 50 mg b.i.d. (Potential Inhibitory Effect of Givinostat on Midazolam IV and on Dabigatran Analysis Population) | 26
Day 7 - Midazolam (Oral) 2.5 mg + Givinostat 50 mg b.i.d. (Potential Inhibitory Effect of Givinostat analysis population) | 26
Days 8-16 - Givinostat 50 mg b.i.d. | 26
Day 17 - Midazolam (IV) 1 mg + Dabigatran 75 mg + Givinostat 50 mg b.i.d. (Potential Inducing Effect of Givinostat on Midazolam IV and on Dabigatran Analysis Population.) | 26
Day 18 - Midazolam (Oral) 2.5 mg + Givinostat 50 mg b.i.d. (Potential Inducing Effect of Givinostat on Oral Midazolam Analysis Population.) | 26
Day 19 - Givinostat 50 mg | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic Analysis Population:Twenty-six (26) subjects were enrolled in Part 1 of the study and provided evaluable pharmacokinetic data for at least one IMP, without deviations affecting pharmacokinetic interpretation.
Groups:
- Number of Subjects Enrolled: Twenty-six (26) subjects (7 women and 19 men) were admitted to study Part 1.
Arm/Group | Number of Subjects Enrolled
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Portugal | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Midazolam, 1-hydroxymidazolam, Following Single Doses of the Parent Drug
Description: Maximum observed plasma concentration (Cmax) of midazolam and 1-hydroxymidazolam following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect) and following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 - Potential Inhibitory Effect, and Day 18 - Potential Inducing Effect).
  13 blood samples were collected at pre-dose and at 2 minutes, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12 and 24 hours after the administration of IV midazolam, on Days 1, 6 and 17, to determine midazolam and 1-hydroxymidazolam plasma concentrations. 11 blood samples were collected at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after the administration of oral midazolam, on Days 2, 7 and 18, to determine midazolam and 1-hydroxymidazolam plasma concentrations.
Time Frame: In the turn of 24 hours after IV midazolam, single dose, administered at day 1,6,17 or after oral midazolam, single dose, administered at days 2, 7 and 18.
Population: PK population: Part 1 Pharmacokinetic Analysis Population includes all subjects enrolled in Part 1 of the study, who provided evaluable pharmacokinetic data for at least one IMP, without deviations affecting pharmacokinetic interpretation.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Groups:
- Midazolam IV Alone (Day 1): A single dose of midazolam 1 mg i.v. was administered on Day 1, 1 hour after givinostat administration.
- Midazolam IV Co-administered With Givinostat (Day 6): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat (at Day 6) to study this latter potential inhibitory effect on midazolam.
  Givinostat 10 mg/mL oral suspension was administered once, in the morning, in Day 6.
- Midazolam IV Co-administered With Givinostat (Day 17): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat (at Day 17) to study this latter potential inducing effect on midazolam.
  Givinostat 10 mg/mL oral suspension was administered once, in the morning, in Day 17.
  Givinostat 10 mg/mL: 10 mg/mL oral suspension. Givinostat 10 mg/ml oral suspension was administered once, in the morning, in Day 17).
- Oral Midazolam Alone (Day 2): A single oral dose of midazolam 2.5 mg oral solution was administered alone.
- Oral Midazolam Co-Administered With Givinostat (Day 7): A single oral dose of midazolam 2.5 mg oral solution was administered, 1 hour after the planned morning time of givinostat administration. The potential Inhibitory Effect of midazolam was assessed
- Oral Midazolam Co-Administered With Givinostat (Day 18): A single oral dose of midazolam 2.5 mg oral solution was administered on day 18, 1 hour after the planned morning time of givinostat administration. The potential inducing effect of midazolam was assessed.
Arm/Group | Midazolam IV Alone (Day 1) | Midazolam IV Co-administered With Givinostat (Day 6) | Midazolam IV Co-administered With Givinostat (Day 17) | Oral Midazolam Alone (Day 2) | Oral Midazolam Co-Administered With Givinostat (Day 7) | Oral Midazolam Co-Administered With Givinostat (Day 18)
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26
pg/mL
  midazolam | 50482.44 [42802.65 to 59540.16] | 53345.17 [46868.39 to 60716.97] | 46510.23 [38309.42 to 56466.57] | 12695.07 [11193.89 to 14397.57] | 15744.30 [13936.13 to 17787.09] | 17678.67 [15782.69 to 19802.43]
  1-hydroxymidazolam | 1426.41 [1269.56 to 1602.64] | 1306.05 [1146.91 to 1487.26] | 1335.02 [1115.15 to 1598.25] | 4451.49 [3756.90 to 5274.51] | 5229.06 [4445.58 to 6150.63] | 6303.67 [5046.18 to 7874.53]
Statistical Analysis 1: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 6); Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV. Cmax; Test type: Other — please note that GMR corresponds to the ratio of the Geometric LSmeans of Midazolam IV Co-Administered with Givinostat (Day 6) and the Geometric LSmeans of Midazolam of IV Alone (Day 1); ratio of the geometric least square mean = 105.67, 90% CI 2-sided [91.72 to 121.74]
Statistical Analysis 2: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 6); 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV - Cmax; Test type: Other — [test comment as in outcome 1, analysis 1]; ratio of the geometric least square mean = 91.56, 90% CI 2-sided [86.16 to 97.31]
Statistical Analysis 3: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 17); Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV - Cmax; Test type: Other — please note that GMR corresponds to the ratio of the Geometric LSmeans of Midazolam IV Co-Administered with Givinostat (Day 17) and the Geometric LSmeans of Midazolam of IV Alone (Day 1); ratio of the Geometric LSmeans = 92.13, 90% CI 2-sided [75.97 to 111.73]
Statistical Analysis 4: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 17); 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV - Cmax; Test type: Other — [test comment as in outcome 1, analysis 3]; ratio of the Geometric LSmeans = 93.59, 90% CI 2-sided [83.72 to 104.63]
Statistical Analysis 5: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 7); Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam - Cmax; Test type: Other — GMR corresponds to the ratio of the Geometric LSmeans of Oral Midazolam Co-Administered with Givinostat (Day 7) and the Geometric LSmeans of Oral Midazolam Alone (Day 2); ratio of the Geometric LSmeans = 124.02, 90% CI 2-sided [114.38 to 134.47]
Statistical Analysis 6: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 7); 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam - Max; Test type: Other — [test comment as in outcome 1, analysis 5]; ratio of the Geometric LSmeans = 117.47, 90% CI 2-sided [104.78 to 131.69]
Statistical Analysis 7: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 18); Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam - Cmax; Test type: Other — GMR corresponds to the ratio of the Geometric LSmeans of Oral Midazolam Co-Administered with Givinostat (Day 18) and the Geometric LSmeans of Oral Midazolam Alone (Day 2); ratio of geometric LS means = 139.28, 90% CI 2-sided [128.71 to 150.67]
Statistical Analysis 8: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 18); 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam - Cmax; Test type: Other — [test comment as in outcome 1, analysis 7]; ratio of geometric LS means = 141.61, 90% CI 2-sided [122.36 to 163.88]

2. Primary Outcome: Cmax for Dabigatran (Total and Free), Following Single Doses of the Parent Drug
Description: Maximum observed plasma concentration (Cmax) of total dabigatran and free dabigatran following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect).
  Fifteen (15) blood samples were collected in K2-EDTA collection tubes at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after the administration of dabigatran etexilate, on Days 1, 6 and 17, for the determination of total and free dabigatran plasma concentrations.
Time Frame: In the turn of 72 hours after administration of dabigatran on day 1,6,17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Dabigatran Etexilate Alone (Day 1): Dabigatran etexilate 75 mg, 1 hard capsule, was administered alone.
- Dabigatran Etexilate Co-Administered With Givinostat (Day 6); Dabigatran Etexilate Co-Administered With Givinostat (Day 17): Dabigatran etexilate 75 mg, 1 hard capsule, was administered 1 hour after the planned morning time of givinostat.
Arm/Group | Dabigatran Etexilate Alone (Day 1) | Dabigatran Etexilate Co-Administered With Givinostat (Day 6) | Dabigatran Etexilate Co-Administered With Givinostat (Day 17)
Number analyzed (Participants) | 26 | 26 | 26
ng/mL
  total dabigatran | 69.44 [51.90 to 92.92] | 51.17 [39.62 to 66.08] | 45.35 [34.87 to 58.99]
  free dabigatran | 60.19 [44.64 to 81.14] | 44.03 [34.49 to 56.21] | 37.41 [29.01 to 48.23]
Statistical Analysis 1: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 6); Total Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - Cmax; Test type: Other — GMR corresponds to the ratio of the Geometric LSmeans of Dabigatran Etexilate Co-Administered with Givinostat (Day 6) and the Geometric LSmeans of Dabigatran Etexilate Alone (Day 1); ratio of the Geometric LSmeans = 73.68, 90% CI 2-sided [60.77 to 89.33]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 6); Free Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - Cmax; Test type: Other — [test comment as in outcome 2, analysis 1]; ratio of the Geometric LSmeans = 70.38, 90% CI 2-sided [57.94 to 85.50]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 17); Total Dabigatran: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - Cmax; Test type: Other — GMR corresponds to the ratio of the Geometric LSmeans of Dabigatran Etexilate Co-Administered with Givinostat (Day 17) and the Geometric LSmeans of Dabigatran Etexilate Alone (Day 1); ratio of the Geometric LSmeans = 65.31, 90% CI 2-sided [53.33 to 79.98]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 17); Free Dabigatran: Potential Induction Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate. Cmax; Test type: Other — [test comment as in outcome 2, analysis 3]; ratio of the Geometric LSmeans = 62.18, 90% CI 2-sided [50.86 to 75.95]

3. Primary Outcome: Tmax for Midazolam, 1-hydroxymidazolam, Following Single Doses of the Parent Drug
Description: tmax =Time of occurrence of Cmax. 13 blood samples were collected at pre-dose and at 2 minutes, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12 and 24 hours after the administration of IV midazolam, on Days 1, 6 and 17, to determine midazolam and 1-hydroxymidazolam plasma concentrations. 11 blood samples were collected at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after the administration of oral midazolam, on Days 2, 7 and 18, to determine midazolam and 1-hydroxymidazolam plasma concentrations.
Time Frame: as for outcome 1
Population: PK population: Part 1 Pharmacokinetic Analysis Population includes all subjects enrolled in Part 1 of the study, who provided evaluable pharmacokinetic data for at least one IMP,
Measure: Median (Full Range); unit: hours
Groups:
- Midazolam IV Alone (Day 1): A single dose of midazolam 1 mg i.v. was administered on Day 1, 1 hour after givinostat administration.
  Midazolam (and dabigatran etexilate) was administered with the subjects in a semi-recumbent position. Subjects remained semirecumbent until at least 3 hours post-dose.
- Midazolam IV Co-administered With Givinostat (Day 17): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat (at Day 17) to study this latter potential inducing effect on midazolam.
  Givinostat 10 mg/mL oral suspension was administered once, in the morning, in Day 17.
- Oral Midazolam Co-Administered With Givinostat (Day 7); Oral Midazolam Co-Administered With Givinostat (Day 18): A single oral dose of midazolam 2.5 mg oral solution was administered.
Arm/Group | Midazolam IV Alone (Day 1) | Midazolam IV Co-administered With Givinostat (Day 6) | Midazolam IV Co-administered With Givinostat (Day 17) | Oral Midazolam Alone (Day 2) | Oral Midazolam Co-Administered With Givinostat (Day 7) | Oral Midazolam Co-Administered With Givinostat (Day 18)
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26
hours
  midazolam | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.25] | 0.55 [0.50 to 1.50] | 0.50 [0.50 to 1.50] | 0.50 [0.50 to 1.02]
  1-hydroxymidazolam | 0.50 [0.25 to 1.00] | 0.50 [0.25 to 2.00] | 0.51 [0.25 to 2.00] | 0.55 [0.50 to 1.50] | 0.50 [0.50 to 1.50] | 0.50 [0.50 to 1.02]

4. Primary Outcome: Tmax for Dabigatran (Total and Free), Following Single Doses of the Parent Drug
Description: The time of occurrence of maximum observed concentration (tmax) of total dabigatran and free dabigatran following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect).
  Fifteen (15) blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after the administration of dabigatran etexilate, on Days 1, 6 and 17, for the determination of total and free dabigatran plasma concentrations.
Time Frame: In the turn of 72 hours after administration of dabigatran on day 1,6,17
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Groups:
- Dabigatran Etexilate Co-Administered With Givinostat (Day 6): Dabigatran etexilate 75 mg, 1 hard capsule, was administered 1 hour after the planned morning time of givinostat administration The Potential Inhibitory Effect on day 6 was assessed.
- Dabigatran Etexilate Co-Administered With Givinostat (Day 17): Dabigatran etexilate 75 mg, 1 hard capsule, was administered. The Potential inducing Effect on day 17 was assessed.
Arm/Group | Dabigatran Etexilate Alone (Day 1) | Dabigatran Etexilate Co-Administered With Givinostat (Day 6) | Dabigatran Etexilate Co-Administered With Givinostat (Day 17)
Number analyzed (Participants) | 26 | 26 | 26
hours
  total dabigatran | 2.00 [1.50 to 4.00] | 2.00 [1.00 to 4.02] | 2.00 [1.00 to 4.00]
  free dabigatran | 2.00 [1.00 to 4.00] | 2.00 [1.50 to 4.02] | 2.00 [1.50 to 6.00]

5. Primary Outcome: t1/2 of Midazolam, 1-hydroxymidazolam, Following Single Doses of Givinostat
Description: T1/2 is the Apparent terminal elimination half-life, calculated as ln(2)/λz. t1/2 of midazolam and 1-hydroxymidazolam following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect) and following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 - Potential Inhibitory Effect, and Day 18 - Potential Inducing Effect).
  13 blood samples were collected at pre-dose and at 2 minutes, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12 and 24 hours after the administration of IV midazolam, on Days 1, 6 and 17, to determine midazolam and 1-hydroxymidazolam plasma concentrations. 11 blood samples were collected at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after the administration of oral midazolam, on Days 2, 7 and 18, to determine midazolam and 1-hydroxymidazolam plasma concentrations.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis includes all subjects enrolled in Part 1 who provided evaluable pk data for at least one IMP. These were: n=26 for (1-Hydroxy)midazolam IV alone, n=25 for (1-Hydroxy)midazolam + givinostat at day 6, n=23 for (1-Hydroxy)midazolam + givinostat at day 17, n=25 for oral (1-Hydroxy)midazolam alone at day 2, n=25 for oral (1-Hydroxy)midazolam + givinostat at day 18 , n=26 for oral midazolam + givinostat at day 7, n=24 for oral 1-Hydroxymidazolam + givinostat at day 7.
Measure: Mean (Full Range); unit: hours
Groups:
- Midazolam IV Alone (Day 1): A single dose of midazolam 1 mg i.v. was administered.
- Midazolam IV Co-administered With Givinostat (Day 6): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat Givinostat 10 mg/mL oral suspension was administered once, in the morning in Day 6.
- Midazolam IV Co-administered With Givinostat (Day 17): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat to study this latter potential inducing effect on midazolam.
  From the Day 4 to Day 18, Givinostat oral suspension (50 mg) was administered twice a day, in the morning and in the evening.
- Oral Midazolam Co-Administered With Givinostat (Day 7): A single oral dose of midazolam 2.5 mg oral solution was administered. The potential Inhibitory Effect of midazolam was assessed .
- Oral Midazolam Co-Administered With Givinostat (Day 18): A single oral dose of midazolam 2.5 mg oral solution was administered. The potential inducing effect of midazolam was assessed.
Arm/Group | Midazolam IV Alone (Day 1) | Midazolam IV Co-administered With Givinostat (Day 6) | Midazolam IV Co-administered With Givinostat (Day 17) | Oral Midazolam Alone (Day 2) | Oral Midazolam Co-Administered With Givinostat (Day 7) | Oral Midazolam Co-Administered With Givinostat (Day 18)
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26
hours
  midazolam: number analyzed (Participants) | 26 | 25 | 23 | 25 | 26 | 25
  midazolam | 5.27 [4.60 to 6.04] | 5.22 [4.61 to 5.90] | 6.62 [5.83 to 7.51] | 5.48 [4.75 to 6.32] | 5.84 [5.08 to 6.70] | 6.73 [5.89 to 7.70]
  1-hydroxymidazolam: number analyzed (Participants) | 26 | 25 | 23 | 25 | 24 | 25
  1-hydroxymidazolam | 4.02 [3.41 to 4.74] | 5.00 [4.20 to 5.95] | 5.74 [4.70 to 7.03] | 4.62 [3.63 to 5.89] | 6.09 [4.76 to 7.80] | 6.43 [5.16 to 8.01]

6. Primary Outcome: t1/2 for Dabigatran (Total and Free), Following Single Doses of the Parent Drug
Description: Apparent terminal elimination half-life, calculated as ln(2)/λz. The t1/2 of total dabigatran and free dabigatran following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect).
  Fifteen (15) blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after the administration of dabigatran etexilate, on Days 1, 6 and 17, for the determination of total and free dabigatran plasma concentrations.
Time Frame: In the turn of 72 hours after administration of dabigatran on day 1,6,17
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Groups:
- Dabigatran Etexilate Co-Administered With Givinostat (Day 6): Dabigatran etexilate 75 mg, 1 hard capsule, was administered 1 hour after the planned morning time of givinostat. The Potential Inhibitory Effect on day 6 was assessed.
- Dabigatran Etexilate Co-Administered With Givinostat (Day 17): Dabigatran etexilate 75 mg, 1 hard capsule, was administered 1 hour after the planned morning time of givinostat administration. The Potential inducing Effect on day 17 was assessed.
Arm/Group | Dabigatran Etexilate Alone (Day 1) | Dabigatran Etexilate Co-Administered With Givinostat (Day 6) | Dabigatran Etexilate Co-Administered With Givinostat (Day 17)
Number analyzed (Participants) | 26 | 26 | 26
hours
  total dabigatran | 7.96 [7.52 to 8.42] | 8.01 [7.21 to 8.90] | 8.74 [8.17 to 9.36]
  free dabigatran: number analyzed (Participants) | 26 | 26 | 25
  free dabigatran | 7.28 [6.73 to 7.89] | 7.03 [6.35 to 7.77] | 8.05 [7.30 to 8.88]

7. Primary Outcome: AUC0-t of Midazolam, 1-hydroxymidazolam, Following Single Doses of Givinostat
Description: AUC0-t =area under the curve from time zero to last sampling time with quantifiable concentrations. AUC0-t of midazolam and 1-hydroxymidazolam following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect) and following Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 - Potential Inhibitory Effect, and Day 18 - Potential Inducing Effect).
  13 blood samples were collected at pre-dose and at 2 minutes, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12 and 24 hours after the administration of IV midazolam, on Days 1, 6 and 17, to determine midazolam and 1-hydroxymidazolam plasma concentrations. 11 blood samples were collected at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after the administration of oral midazolam, on Days 2, 7 and 18, to determine midazolam and 1-hydroxymidazolam plasma concentrations.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: pg.h/mL
Groups:
- Midazolam IV Alone (Day 1): A single dose of midazolam 1 mg i.v. was administered on Day 1. Midazolam (and dabigatran etexilate) was administered with the subjects in a semi-recumbent position. Subjects remained semirecumbent until at least 3 hours post-dose.
- Midazolam IV Co-administered With Givinostat (Day 6): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat (at Day 6) to study this latter potential inhibitory effect on midazolam.
- Midazolam IV Co-administered With Givinostat (Day 17): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat (at Day 17) to study this latter potential inducing effect on midazolam.
- Oral Midazolam Co-Administered With Givinostat (Day 7): A single oral dose of midazolam 2.5 mg oral solution was administered on day 7, 1 hour after the planned morning time of givinostat administration. The potential Inhibitory Effect of midazolam was assessed (day 7)
- Oral Midazolam Co-Administered With Givinostat (Day 18): A single oral dose of midazolam 2.5 mg oral solution was administered on day 18, 1 hour after the planned morning time of givinostat administration. The potential inducing effect of midazolam was assessed (day 18)
Arm/Group | Midazolam IV Alone (Day 1) | Midazolam IV Co-administered With Givinostat (Day 6) | Midazolam IV Co-administered With Givinostat (Day 17) | Oral Midazolam Alone (Day 2) | Oral Midazolam Co-Administered With Givinostat (Day 7) | Oral Midazolam Co-Administered With Givinostat (Day 18)
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26
pg.h/mL
  Midazolam | 44094.42 [39998.55 to 48609.70] | 47333.50 [43297.80 to 51745.35] | 53692.16 [48609.52 to 59306.23] | 36483.20 [31064.96 to 42846.48] | 50134.44 [42444.64 to 59217.42] | 57559.53 [49279.79 to 67230.40]
  1-hydroxymidazolam | 5050.60 [4441.81 to 5742.83] | 5362.65 [4757.51 to 6044.76] | 6210.86 [5374.62 to 7177.22] | 10871.00 [9475.99 to 12471.38] | 14264.35 [12357.51 to 16465.42] | 17208.29 [14624.58 to 20248.46]
Statistical Analysis 1: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 6); Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV - AUC0-t; Test type: Other — GMR corresponds to the ratio of the Geometric LSmeans of Midazolam IV Co-Administered with Givinostat (Day 6) and the Geometric LSmeans of Midazolam of IV Alone (Day 1); ratio of the geometric LS means = 107.35, 90% CI 2-sided [103.35 to 111.49]
Statistical Analysis 2: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 6); 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV - AUC0-t; Test type: Other — [test comment as in outcome 7, analysis 1]; ratio of the Geometric LSmeans = 106.18, 90% CI 2-sided [100.84 to 111.80]
Statistical Analysis 3: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 17); Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV - AUC0-t; Test type: Other — GMR corresponds to the ratio of the Geometric LSmeans of Midazolam IV Co-Administered with Givinostat (Day 17) and the Geometric LSmeans of Midazolam of IV Alone (Day 1); ratio of the Geometric LSmeans = 121.77, 90% CI 2-sided [117.56 to 126.12]
Statistical Analysis 4: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 17); 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV - AUC0-t; Test type: Other — [test comment as in outcome 7, analysis 3]; ratio of the Geometric LSmeans = 122.97, 90% CI 2-sided [115.08 to 131.41]
Statistical Analysis 5: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 7); Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam - AUC0-t; Test type: Other — [test comment as in outcome 1, analysis 5]; ratio of the Geometric LSmeans = 137.42, 90% CI 2-sided [128.09 to 147.43]
Statistical Analysis 6: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 7); 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam - AUC0-t; Test type: Other — [test comment as in outcome 1, analysis 5]; ratio of the Geometric LSmeans = 131.21, 90% CI 2-sided [122.47 to 140.59]
Statistical Analysis 7: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 18); Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam. - AUC0-t; Test type: Other — [test comment as in outcome 1, analysis 7]; ratio of the Geometric LSmeans = 157.77, 90% CI 2-sided [147.49 to 168.76]
Statistical Analysis 8: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 18); 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: - AUC0-t; Test type: Other — [test comment as in outcome 1, analysis 7]; ratio of the Geometric LSmeans = 158.30, 90% CI 2-sided [145.23 to 172.54]

8. Primary Outcome: AUC0-t for Dabigatran (Total and Free), Following Single Doses of the Parent Drug
Description: AUC0-t =area under the curve from time zero to last sampling time with quantifiable concentrations. AUC0-t of total dabigatran and free dabigatran following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect).
  Fifteen (15) blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after the administration of dabigatran etexilate, on Days 1, 6 and 17, for the determination of total and free dabigatran plasma concentrations.
Time Frame: In the turn of 72 hours after administration of dabigatran on day 1,6,17
Population: as for outcome 1
Measure: Median (Full Range); unit: ng.h/mL
Groups:
- Dabigatran Etexilate Co-Administered With Givinostat (Day 6): Dabigatran etexilate 75 mg, 1 hard capsule, was administered 1 hour after the planned morning time of givinostat administration. The Potential Inhibitory Effect on day 6 was assessed.
Arm/Group | Dabigatran Etexilate Alone (Day 1) | Dabigatran Etexilate Co-Administered With Givinostat (Day 6) | Dabigatran Etexilate Co-Administered With Givinostat (Day 17)
Number analyzed (Participants) | 26 | 26 | 26
ng.h/mL
  total dabigatran | 552.25 [424.19 to 718.98] | 386.05 [299.12 to 498.25] | 386.23 [306.46 to 486.78]
  free dabigatran | 460.16 [341.52 to 620.01] | 341.01 [268.24 to 433.52] | 332.71 [268.91 to 411.66]
Statistical Analysis 1: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 6); Total Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics - AUC0-t; Test type: Other — [test comment as in outcome 2, analysis 1]; ratio of the Geometric LSmeans = 69.90, 90% CI 2-sided [58.43 to 83.64]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 6); Free Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - AUC0-t; Test type: Other — [test comment as in outcome 2, analysis 1]; ratio of the Geometric LSmeans = 71.43, 90% CI 2-sided [58.67 to 86.98]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 17); Total Dabigatran: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - AUC0-t; Test type: Other — [test comment as in outcome 2, analysis 3]; ratio of the Geometric LSmeans = 69.94, 90% CI 2-sided [58.82 to 83.15]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 17); Free Dabigatran: Potential Induction Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - AUC0-t; Test type: Other — [test comment as in outcome 2, analysis 3]; ratio of the Geometric LSmeans = 72.30, 90% CI 2-sided [59.92 to 87.25]

9. Primary Outcome: AUC0-inf of Midazolam, 1-hydroxymidazolam, Following Single Doses of Givinostat
Description: AUC0-inf=Total AUC extrapolated to infinity, calculated as AUC0-t + Clast/λz, where Clast is the last measurable concentration and λz is the apparent terminal elimination rate constant.
  13 blood samples were collected at pre-dose and at 2 minutes, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12 and 24 hours after the administration of IV midazolam, on Days 1, 6 and 17, to determine midazolam and 1-hydroxymidazolam plasma concentrations. 11 blood samples were collected at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after the administration of oral midazolam, on Days 2, 7 and 18, to determine midazolam and 1-hydroxymidazolam plasma concentrations.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis includes all subjects enrolled in Part 1 who provided evaluable pk data for at least one IMP. These were:
  n=26 for (1-Hydroxy)midazolam IV alone, n=26 for Mid IV + givinostat (G) at days 6 and 17, for oral hydroxymid alone at day 2, oral Mid + G at day 7.
  n=25 for 1-Hydroxymid + G at day 6, oral mid alone at day 2, oral (1-Hydroxy)mid + G at day 18.
  n=24 for oral 1-Hydroxymid + G at day 7 n=23 for oral 1-hydroxymid + G at day 17
Measure: Median (Full Range); unit: pg.h/mL
Groups:
- Midazolam IV Co-administered With Givinostat (Day 6): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat to study this latter potential inhibitory effect on midazolam.
- Midazolam IV Co-administered With Givinostat (Day 17): Midazolam IV 1 mg/ml, single dose, was co-administered with givinostat to study this latter potential inducing effect on midazolam.
- Oral Midazolam Co-Administered With Givinostat (Day 7): A single oral dose of midazolam 2.5 mg oral solution was administered on day 7, 1 hour after the planned morning time of givinostat administration. The potential Inhibitory Effect of midazolam was assessed.
Arm/Group | Midazolam IV Alone (Day 1) | Midazolam IV Co-administered With Givinostat (Day 6) | Midazolam IV Co-administered With Givinostat (Day 17) | Oral Midazolam Alone (Day 2) | Oral Midazolam Co-Administered With Givinostat (Day 7) | Oral Midazolam Co-Administered With Givinostat (Day 18)
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26
pg.h/mL
  Midazolam: number analyzed (Participants) | 26 | 26 | 26 | 25 | 26 | 25
  Midazolam | 46054.19 [41834.50 to 50699.50] | 49532.66 [45406.00 to 54034.35] | 57112.86 [51342.91 to 63531.25] | 39037.54 [33096.57 to 46044.94] | 53379.48 [45107.58 to 63168.29] | 62904.03 [52906.81 to 74790.32]
  1-Hydroxymidazolam: number analyzed (Participants) | 26 | 25 | 23 | 26 | 24 | 25
  1-Hydroxymidazolam | 5720.13 [4981.56 to 6568.21] | 6404.39 [5615.24 to 7304.43] | 7821.70 [6736.26 to 9082.04] | 11914.16 [10292.86 to 13790.84] | 15895.61 [13769.86 to 18349.51] | 19199.79 [16300.75 to 22614.41]
Statistical Analysis 1: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 6); Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV: AUC0-inf; Test type: Other — [test comment as in outcome 7, analysis 1]; ratio of the Geometric LSmeans = 107.55, 90% CI 2-sided [103.35 to 111.49]
Statistical Analysis 2: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 6); 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV - AUC0-inf; Test type: Other — [test comment as in outcome 7, analysis 1]; ratio of the Geometric LSmeans = 112.17, 90% CI 2-sided [106.21 to 118.46]
Statistical Analysis 3: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 17); Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV - AUC0-inf; Test type: Other — [test comment as in outcome 7, analysis 3]; ratio of the Geometric LSmeans = 124.01, 90% CI 2-sided [119.44 to 128.76]
Statistical Analysis 4: Comparison: Midazolam IV Alone (Day 1) vs Midazolam IV Co-administered With Givinostat (Day 17); 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV. AUC0-inf; Test type: Other — [test comment as in outcome 7, analysis 3]; ratio of the Geometric LSmeans = 134.29, 90% CI 2-sided [126.15 to 142.96]
Statistical Analysis 5: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 7); Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam - AUC0-inf; Test type: Other — [test comment as in outcome 1, analysis 5]; ratio of the Geometric LSmeans = 138.75, 90% CI 2-sided [129.05 to 149.18]
Statistical Analysis 6: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 7); 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: AUC0-inf; Test type: Other; GMR corresponds to the ratio of the Geom = 134.18, 90% CI 2-sided [124.19 to 144.97]
Statistical Analysis 7: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 18); Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: AUC0-inf; Test type: Other — [test comment as in outcome 1, analysis 7]; ratio of the Geometric LSmeans = 162.76, 90% CI 2-sided [151.13 to 175.28]
Statistical Analysis 8: Comparison: Oral Midazolam Alone (Day 2) vs Oral Midazolam Co-Administered With Givinostat (Day 18); 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam - AUC0-inf; Test type: Other — [test comment as in outcome 1, analysis 7]; ratio of the Geometric LSmeans = 161.20, 90% CI 2-sided [147.80 to 175.82]

10. Primary Outcome: AUC0-inf for Dabigatran (Total and Free), Following Single Doses of the Parent Drug
Description: AUC0-inf = Total AUC extrapolated to infinity, calculated as AUC0-t + Clast/λz, where Clast is the last measurable concentration and λz is the apparent terminal elimination rate constant. AUC0-inf of total dabigatran and free dabigatran following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect).
  Fifteen (15) blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after the administration of dabigatran etexilate, on Days 1, 6 and 17, for the determination of total and free dabigatran plasma concentrations.
Time Frame: In the turn of 72 hours after administration of dabigatran on day 1,6,17
Population: as for outcome 1
Measure: Median (Full Range); unit: ng.h/mL
Groups:
- Dabigatran Etexilate Co-Administered With Givinostat (Day 6): Dabigatran etexilate 75 mg, 1 hard capsule, was administered 1 hour after the planned morning time of givinostat administration. The Potential Inhibitory Effect was assessed.
- Dabigatran Etexilate Co-Administered With Givinostat (Day 17): Dabigatran etexilate 75 mg, 1 hard capsule, was administered 1 hour after the planned morning time of givinostat administration. The Potential inducing Effect was assessed.
Arm/Group | Dabigatran Etexilate Alone (Day 1) | Dabigatran Etexilate Co-Administered With Givinostat (Day 6) | Dabigatran Etexilate Co-Administered With Givinostat (Day 17)
Number analyzed (Participants) | 26 | 26 | 26
ng.h/mL
  total dabigatran | 563.09 [436.43 to 726.51] | 393.93 [306.01 to 507.11] | 396.25 [315.23 to 498.10]
  free dabigatran: number analyzed (Participants) | 26 | 26 | 25
  free dabigatran | 467.79 [349.48 to 626.16] | 347.56 [273.95 to 440.95] | 347.73 [280.67 to 430.81]
Statistical Analysis 1: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 6); Total Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - AUC0-inf; Test type: Other — [test comment as in outcome 2, analysis 1]; ratio of the Geometric LSmeans = 69.96, 90% CI 2-sided [58.83 to 83.20]
Statistical Analysis 2: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 6); Free Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - AUC0-inf; Test type: Other — [test comment as in outcome 2, analysis 1]; ratio of the Geometric LSmeans = 71.65, 90% CI 2-sided [59.08 to 86.88]
Statistical Analysis 3: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 17); Total Dabigatran: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate - AUC0-inf; Test type: Other — [test comment as in outcome 2, analysis 3]; ratio of the Geometric LSmeans = 70.37, 90% CI 2-sided [59.64 to 83.03]
Statistical Analysis 4: Comparison: Dabigatran Etexilate Alone (Day 1) vs Dabigatran Etexilate Co-Administered With Givinostat (Day 17); Free Dabigatran: Potential Induction Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate. AUC0-inf; Test type: Other — [test comment as in outcome 2, analysis 3]; ratio of the Geometric LSmeans = 73.45, 90% CI 2-sided [60.79 to 88.75]

11. Primary Outcome: %AUCextrap of Midazolam, 1-hydroxymidazolam, Following Single Doses of Givinostat
Description: Area under the curve or AUC is a pharmacokinetic statistic used to describe the total exposure to a drug. More specifically, it is the time-averaged concentration of drug circulating in the body fluid analyzed (normally plasma, blood or serum). Standard calculation of AUC involves using non-compartmental techniques to calculate the AUC from time 0 to the last measurable concentration. This is called AUC0-t and represents the observed exposure to a drug. The total AUC or AUC0-∞ is the area under the curve from time 0 extrapolated to infinite time.
  %AUCextrap = Percentage of AUC0-∞ due to extrapolation from the time of the last measurable concentration (tlast) to infinity, i.e., residual area, calculated as 100 ∙(AUC0-∞ - AUC0-t) / AUC0-∞.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Percentage of AUC0-inf
Arm/Group | Midazolam IV Alone (Day 1) | Midazolam IV Co-administered With Givinostat (Day 6) | Midazolam IV Co-administered With Givinostat (Day 17) | Oral Midazolam Alone (Day 2) | Oral Midazolam Co-Administered With Givinostat (Day 7) | Oral Midazolam Co-Administered With Givinostat (Day 18)
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26
Percentage of AUC0-inf
  Midazolam: number analyzed (Participants) | 26 | 26 | 26 | 25 | 26 | 25
  Midazolam | 3.87 [3.23 to 4.63] | 3.96 [3.27 to 4.81] | 5.12 [4.07 to 6.43] | 5.02 [4.28 to 5.90] | 5.33 [4.31 to 6.59] | 5.79 [4.46 to 7.52]
  1-Hydroxymidazolam: number analyzed (Participants) | 26 | 25 | 23 | 26 | 26 | 26
  1-Hydroxymidazolam | 9.72 [7.55 to 12.52] | 13.20 [10.09 to 17.27] | 15.97 [12.14 to 21.02] | 6.95 [5.18 to 9.33] | 8.42 [6.62 to 10.70] | 8.80 [7.42 to 10.44]

12. Primary Outcome: %AUC0extrap (%) for Dabigatran (Total and Free), Following Single Doses of the Parent Drug
Description: Area under the curve (AUC) is a pharmacokinetic statistic used to describe the total exposure to a drug. More specifically, it is the time-averaged concentration of drug circulating in the body fluid analyzed. The total AUC (AUC0-∞) is the area under the curve from time 0 extrapolated to infinite time.
  * AUC0extrap = Percentage of AUC0-∞ due to extrapolation from the time of the last measurable concentration (tlast) to infinity, i.e., residual area, calculated as 100 ∙(AUC0-∞ - AUC0-t) / AUC0-∞.
  * AUC0extrap of total dabigatran and free dabigatran following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 - Potential Inhibitory Effect, and Day 17 - Potential Inducing Effect).
  Fifteen (15) blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after the administration of dabigatran etexilate, on Days 1, 6 and 17, for the determination of total and free dabigatra
Time Frame: In the turn of 72 hours after administration of dabigatran on day 1,6,17
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage of AUC0-inf
Arm/Group | Dabigatran Etexilate Alone (Day 1) | Dabigatran Etexilate Co-Administered With Givinostat (Day 6) | Dabigatran Etexilate Co-Administered With Givinostat (Day 17)
Number analyzed (Participants) | 26 | 26 | 26
Percentage of AUC0-inf
  total dabigatran | 1.37 [1.04 to 1.80] | 1.79 [1.50 to 2.15] | 2.23 [1.84 to 2.70]
  free dabigatran: number analyzed (Participants) | 26 | 26 | 25
  free dabigatran | 1.27 [1.00 to 1.62] | 1.69 [1.39 to 2.05] | 2.02 [1.58 to 2.58]

13. Primary Outcome: λz of Midazolam, 1-hydroxymidazolam, Following Single Doses of Givinostat
Description: Apparent first order elimination rate constant associated with the terminal (log-linear) portion of the concentration versus time curve. The parameter is estimated by linear least square regression analysis using the last three (or more) non-zero concentrations.
  13 blood samples were collected at pre-dose and at 2 minutes, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12 and 24 hours after the administration of IV midazolam, on Days 1, 6 and 17, to determine midazolam and 1-hydroxymidazolam plasma concentrations. 11 blood samples were collected at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after the administration of oral midazolam, on Days 2, 7 and 18, to determine midazolam and 1-hydroxymidazolam plasma concentrations.
Time Frame: as for outcome 1
Population: Pharmacokinetic Analysis includes all subjects enrolled in Part 1 who provided evaluable pk data for at least one IMP. These were:
  n=26 for (1-Hydroxy)midazolam IV alone, n=26 for Mid IV + givinostat (G) at days 6 and 17, for oral hydroxymid alone at day 2, oral Mid + G at day 7.
  n=25 for 1-Hydroxymid + G at day 6, oral mid alone at day 2, oral (1-Hydroxy)mid + G at day 18.
  n=24 for oral 1-Hydroxymid + G at day 7 n=23 for IV 1-hydroxymid + G at day 17
Measure: Median (Full Range); unit: 1/h
Arm/Group | Midazolam IV Alone (Day 1) | Midazolam IV Co-administered With Givinostat (Day 6) | Midazolam IV Co-administered With Givinostat (Day 17) | Oral Midazolam Alone (Day 2) | Oral Midazolam Co-Administered With Givinostat (Day 7) | Oral Midazolam Co-Administered With Givinostat (Day 18)
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26 | 26
1/h
  Midazolam: number analyzed (Participants) | 26 | 26 | 26 | 25 | 26 | 25
  Midazolam | 0.131 [0.115 to 0.151] | 0.133 [0.118 to 0.150] | 0.105 [0.092 to 0.119] | 0.127 [0.110 to 0.146] | 0.119 [0.103 to 0.136] | 0.103 [0.090 to 0.118]
  1-Hydroxymidazolam: number analyzed (Participants) | 26 | 25 | 23 | 26 | 24 | 25
  1-Hydroxymidazolam | 0.172 [0.146 to 0.203] | 0.139 [0.116 to 0.165] | 0.121 [0.099 to 0.148] | 0.150 [0.118 to 0.191] | 0.114 [0.089 to 0.146] | 0.108 [0.087 to 0.134]

14. Primary Outcome: λz of Dabigatran (Total and Free), Following Single Doses of Givinostat
Description: Apparent first order elimination rate constant associated with the terminal (log-linear) portion of the concentration versus time curve. The parameter is estimated by linear least square regression analysis using the last three (or more) non-zero concentrations.
  Fifteen (15) blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after the administration of dabigatran etexilate, on Days 1, 6 and 17, for the determination of total and free dabigatran plasma concentrations.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: 1/h
Arm/Group | Dabigatran Etexilate Alone (Day 1) | Dabigatran Etexilate Co-Administered With Givinostat (Day 6) | Dabigatran Etexilate Co-Administered With Givinostat (Day 17)
Number analyzed (Participants) | 26 | 26 | 26
1/h
  Total Dabigatran | 0.087 [0.082 to 0.092] | 0.087 [0.078 to 0.096] | 0.079 [0.074 to 0.085]
  Free dabigatran: number analyzed (Participants) | 26 | 26 | 25
  Free dabigatran | 0.095 [0.088 to 0.103] | 0.099 [0.089 to 0.109] | 0.086 [0.078 to 0.095]

15. Secondary Outcome: Number of Adverse Events by Severity (Mild, Moderate, Severe)
Description: An AE was considered as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily imply a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  The period of observation for the collection of medical occurrences extended from the time when the subject gave Informed Consent until the follow-up visit.
Time Frame: Throughout the study and 10-14 days after the EoS (follow-up visit), i.e. up to date 30-34
Population: All subjects who receive at least one dose of an IMP in Part 1 of the study constitute the Part 1 Safety Analysis Population.
Measure: Number; unit: number of TEAE
Groups:
- Midazolam: Oral or IV, alone or in combination
- Dabigatran: Dabigatran etexilate 75 mg oral hard capsules in combination with Midazolam
- Givinostat: ITF2357/Givinostat* 10 mg/mL oral suspension
- Total: 26 participants overall, despite the Investigational Products Dose and Mode of Administration
Arm/Group | Midazolam | Dabigatran | Givinostat | Total
Number analyzed (Participants) | 26 | 26 | 26 | 26
number of TEAE
  AE mild severity | 28 | 25 | 74 | 127
  AE moderate severity | 0 | 0 | 2 | 2
  AE severe | 0 | 0 | 0 | 0

16. Secondary Outcome: Incidence of Patients With at Least One Adverse Events by Severity (Mild, Moderate, Severe)
Description: as for outcome 15
Time Frame: During the study and 10-14 days after the EoS (follow-up visit), i.e. up to day 30-34
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Dabigatran | Givinostat | Total
Number analyzed (Participants) | 26 | 26 | 26 | 26
Participants
  AE mild severity | 26 | 26 | 26 | 26
  AE moderate severity | 2 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Throughout the study and 10-14 days after the End of Study (safety follow-up visit), i.e. up to day 30-34, all TEAEs, considered related or not related to IMPs, were collected.
Description: End-of-study was defined as the last study procedure on Day 11 or at early discontinuation of subjects administered at least one dose of investigational product.
  Early termination procedures were performed as soon as possible after subject withdrawal, within 10-14 days after last participation of the subject in the study, whenever possible
Groups:
- Midazolam: Midazolam 1mg/ml IV, single dose, was administered on Days 1, 6 and 17, 1 hour after the planned morning time of givinostat administration. Midazolam 2.5 mg single oromucosal solution was administered on Days 2, 7 and 18, 1 hour after the planned morning time of givinostat administration.
- Dabigatran: Dabigatran etexilate 75 mg oral hard capsules Dose: 75 mg; Dosage form: hard capsules On Days 1, 6 and 17, dabigatran etexilate 75 mg was administered (with midazolam 1mg IV) 1 hour after the planned morning time of givinostat administration.
- Givinostat: 10 mg/mL oral suspension. Givinostat 10 mg/ml oral suspension was administered once, in the morning, in Days 1, 2, 6, 7, 17 and 18), and twice a day (50 mg as oral suspension), in the morning and in the evening, from the Day 4 to Day 18. On Day 19, only the morning dose was administered.
Arm/Group | Midazolam | Dabigatran | Givinostat
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 26/26 | 26/26 | 26/26
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=26) | Dabigatran (N=26) | Givinostat (N=26)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (20) | 19 (20) | 19 (20)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 2 (2) | 2 (2) | 2 (2)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 7 (8) | 7 (8)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Faeces soft (Gastrointestinal disorders) | 5 (7) | 5 (7) | 4 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 5 (5)
Oesophageal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 3 (3) | 3 (3)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Transaminases increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 1 (2) | 1 (2) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 17 (35) | 17 (35) | 17 (25)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10) | 10 (10) | 9 (9)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT05492318/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT05492318/SAP_001.pdf